CLINICAL TRIAL: NCT02641600
Title: Randomised Trial Comparing the Effectiveness of Elastic Compression in Treating Chronic Venous Disease (CEAP C2-C5)
Brief Title: Elastic Compression in Chronic Venous Disease
Acronym: RECVEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Stavros Kakkos, Assistant Professor of Vascular Surgery, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35/18.02.2015
Record Dates: First submitted 2015-12-21; First posted 2015-12-29 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Varicosity
MeSH Terms: conditions — Varicose Veins | interventions — Stockings, Compression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elastic stockings (Active Comparator): Class 1 elastic stockings (18-21 mmHg)
  Interventions: Device: Elastic stockings
- Placebo stockings (Placebo Comparator): Placebo stockings (0 mmHg)
  Interventions: Device: Placebo stockings

INTERVENTIONS:
Device: Elastic stockings — Use of elastic stockings to alleviate patient symptoms
  Arms: Elastic stockings
Device: Placebo stockings — Placebo stocking with pressure applied to the legs
  Arms: Placebo stockings

SUMMARY:
Patients with chronic venous disease causing pain or ache will be randomised into two groups, active stockings (18-21 mmHg) or placebo stockings

DETAILED DESCRIPTION:
Patients with chronic venous disease causing pain or ache satisfying the inclusion and exclusion criteria will be randomised into two groups, active stockings (18-21 mmHg) or placebo stockings. The primary outcome of the study (pain/ache scored using a visual analogue scale) and a number of secondary symptoms, signs and rVCSS (revised Venous Clinical Severity Score) will be obtained at baseline and after one week of wearing the active or placebo stocking.

ELIGIBILITY:
Inclusion Criteria:

* Primary varicose veins causing pain/ache located only at the calf level

Exclusion Criteria:

* Venous ulceration
* Dermatitis
* Itching
* Superficial vein thrombosis
* Peripheral arterial disease
* Symptoms of non-venous origin
* Previous use of elastic stockings

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Pain/ache assessed using a visual analogue scale (0-10) | One week
  Patients with varicose veins often complain for dull pain of ache. This will be assessed using a visual analogue scale (0-10)

SECONDARY OUTCOMES:
revised Venous Clinical Severity Score (rVCSS) | One week
  revised Venous Clinical Severity Score
Heaviness assessed using a visual analogue scale (0-10) | One week
  Patients with varicose veins often complain for heaviness. This will be assessed using a visual analogue scale (0-10)
Night cramps assessed using a visual analogue scale (0-10) | One week
  Patients with varicose veins often complain for night cramps. These will be assessed using a visual analogue scale (0-10)
Swelling sensation assessed using a visual analogue scale (0-10) | One week
  Patients with varicose veins often complain for sensation of swelling. This will be assessed using a visual analogue scale (0-10)
Burning sensation assessed using a visual analogue scale (0-10) | One week
  Patients with varicose veins often complain for burning sensation. This will be assessed using a visual analogue scale (0-10)
Paresthesia assessed using a visual analogue scale (0-10) | One week
  Patients with varicose veins often complain for paresthesia. This will be assessed using a visual analogue scale (0-10)
Restless legs assessed using a visual analogue scale (0-10) | One week
  Patients with varicose veins often complain for restless legs. This symptom will be assessed using a visual analogue scale (0-10)
throbbing assessed using a visual analogue scale (0-10) | One week
  Patients with varicose veins often complain for throbbing of their varicose veins. This will be assessed using a visual analogue scale (0-10)
insomnia assessed using a visual analogue scale (0-10) | One week
  Patients with varicose veins often complain for insomnia. This will be assessed using a visual analogue scale (0-10)
Ankle circumference | One week
  This will be measured just above the malleoli, at the smallest point.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros K Kakkos, MD, PhD, Principal Investigator — University of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece